CLINICAL TRIAL: NCT05986539
Title: Mechanistic Effects of Early Life Feeding Exposure on Infant Inflammatory and Health Status
Brief Title: Early Life Feeding Exposure and Infant Immune and Health Status.
Status: Recruiting | Type: Observational
Sponsor: University of Idaho (Other)
Responsible Party: Principal Investigator, Bethaney Fehrenkamp, Clinical Assistant Professor, University of Idaho
Other Study IDs: 23-013
Record Dates: First submitted 2023-06-21; First posted 2023-08-14 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Maternal Behavior; Maternal Obesity; Breast Milk Collection; Infant Development
MeSH Terms: conditions — Pregnancy in Obesity; Breast Milk Expression | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breastmilk samples will be collected when a woman is breastfeeding. Infant fecal samples will be collected. Maternal and infant blood samples will be collected. Women can optionally submit saliva and fecal samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breastfeeding dyad: Women, and their infants, that intend to exclusively breastfeed or begin using formula as supplemental to breastmilk throughout the study.
  Interventions: Other: Observational
- Formula feeding dyads: Women, and their infants, that intend to exclusively use formula from 6-18 weeks of life, the duration of the study,
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This study is only observational in nature and will not include an intervention.
  Other Names: Observation only based on natural experiment of feeding groups

SUMMARY:
Background: Although breastfeeding has known protective effects, such as preventing childhood obesity, the specific mechanisms remain unclear. Idaho has a high breastfeeding initiation rate (92%) but a significant prevalence of childhood obesity (30.5% overweight/obese). Limited research exists on the impact of maternal inflammation, maternal body mass index (BMI), C-reactive protein (CRP), and interleukin-6 (IL-6) concentrations in breastmilk on infant health outcomes, especially in healthy full-term infants.

Objective: This study aims to expand understanding of the role of maternal inflammation on breastmilk composition and its effect on infant immune development. The investigators seek to investigate the relationship between maternal health status, breastmilk inflammatory concentrations, and balanced immune development in infants. Additionally, the investigators aim to explore the potential influence of early diet exposure, including maternal inflammatory status, on the risk of obesity and other inflammatory conditions.

Methods: Healthy full-term infants (breastfed/formula-fed) and their mothers will be recruited. Maternal inflammation markers (BMI, CRP, IL-6) and immune markers in infants will be analyzed. Flow cytometry will assess immune populations. Correlations between maternal systemic inflammation, infant inflammation, and breastmilk inflammatory markers will be examined for breastfeeding mothers.

Outcomes: The investigators hypothesize breastfed infants will display a more favorable anti-inflammatory profile. This study will identify factors influencing immune development and potential pathways linking early-life exposures to long-term health outcomes. Findings will inform strategies for promoting balanced immune development and elucidate the role of early diet exposure, including maternal inflammation, as a protective or risk factor for obesity and inflammatory conditions.

DETAILED DESCRIPTION:
The immune system of newborns is immature and undergoes rapid development during the first few months of life. Inflammation is a natural response to infection or tissue injury, but excessive or prolonged inflammation can be detrimental to immune development. Understanding the relationship between inflammation and immune development in healthy full-term infants is critical to developing effective interventions to promote healthy immune function in early life.

This project will collect blood samples from healthy full-term infants at 2 and 4 months of age. The samples will be analyzed using flow cytometry to quantify the proportions and activation status of different immune cell populations, such as T, B, natural killer, and monocytes. The analysis will also include quantifying intracellular cytokines to assess the functional capacity of the immune cells. The samples will be analyzed using established methods to measure biomarkers of inflammation, such as CRP, TNF-alpha, and other inflammatory interleukins and cytokines. This project will expand upon biomarkers previously examined to aid in the overall understanding of the role of inflammation in healthy immune development. Fecal samples will be collected from infants five times during the first 6 to 18 weeks of life. Fecal CRP and calprotectin levels will be quantified to detect low-level inflammation and enhance systemic results. Breastmilk will also be collected from lactating women at corresponding collection times to assess breastfeeding's impact on immune development. In addition to data collected on maternal BMI, maternal blood will be collected at 2 and 4 months postpartum to enhance investigations into maternal inflammatory status. Using existing clinical partnerships, 30 maternal-infant dyads will be recruited during the first 6 weeks of life and followed for 12 weeks. Dyads will include 15 breastfeeding infants, to be matched with 15 infants receiving formula or other non-human-based milk products (i.e., plant based formula). Dyads will be matched on infant sex and maternal BMI. A human milk sample will be collected at 6, 8, 12, 16 and 18 weeks postpartum in connection with infant fecal samples (Figure 1). Mothers can opt-in to collecting their own feces and saliva. Blood will be obtained from infants during recurring pediatric wellness visits. Mothers will also be asked to complete reoccurring surveys regarding their diet, perceived stress and anxiety, infant diet, food introduction, and general infant behavior or level of fussiness. Maternal demographics, including education level, household income, and food security, will be collected upon enrollment. Electronic medical records will be accessed related to prenatal care; maternal health and pre-existing conditions; birth records; and infant health status, including growth and incidence of infection and use of antibiotics. The investigators will measure the concentrations of inflammatory cytokines in fecal and blood samples from infants and in milk and blood samples from their mothers. Flow cytometry will analyze infant and maternal blood samples for circulating immune cell populations. When available, saliva samples will be analyzed for cortisol concentration. Remaining infant and maternal fecal samples will be retained for future microbiome investigations.

ELIGIBILITY:
Inclusion Criteria:

* Mother at least 18 years of age
* Mother is in third trimester (week 27 of gestation) or biological infant is 5 weeks of age or younger
* Mother plans to continue to provide your infant breastmilk (by breastfeeding or by pumping) for at least 18 weeks (4.5 months) from your delivery date or mother plans to continue to provide formula exclusively to infant for at least 18 weeks of life.
* Mother lives within a 45-mile radius of Study Site, or is willing to deliver samples for visits 2, 4, and 6.
* Mother willing to meet at (designated sample collection site) for visits 3 and 5 for sample collection and visit activities.
* Mother willing to consent and comply with all aspects of the study protocol and methods, save the optional activities and optional sample collections.
* Mother and infant are considered healthy by Principle Investigator.
* For Formula Fed Group: Mother-Infant dyad is able to match to a Breastfed dyad using maternal BMI and infant sex.

Exclusion Criteria:

* Mother or Infant have participated or are currently participating in an interventional drug or device (non-observational) research study before.
* Mother reports that they, or the infant, have had an adverse effect during a venous blood collection.
* Infant was born less than 36 weeks of gestation.
* Infant or mother have health conditions that increase the risk of study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This project is focused on the effects of maternal inflammation and health status on the developing infant, including the role of breastfeeding and early feeding practices.
Study Population: Study population is postnatal women and their infant dyads.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Characterize the change in systemic inflammatory profile of healthy full-term infants | Through study completion, an average of 12 weeks.
  We will investigate infant inflammation across the first 4.5 months of life in serum and feces using biomarkers C-reactive protein, tumor necrosis factor-alpha, and other inflammatory interleukins and cytokines.

SECONDARY OUTCOMES:
Characterize the potential correlation between maternal systemic inflammation and inflammatory profile of the breastmilk. | Through study completion, an average of 12 weeks.
  We will explore how maternal systemic inflammation may correlate with inflammatory markers within the breastmilk. We hypothesize that maternal systemic inflammation and health status will be correlated with increased inflammatory markers in breast milk if breastfeeding.

OTHER OUTCOMES:
Characterize the change in blood mononuclear cell distribution of healthy full term infants. | Through study completion, an average of 12 weeks.
  We will assess this relationship by flow cytometry analysis of peripheral blood mononuclear cells at 2 and 4 months of age. We expect to capture biological variation in circulating immune cell populations in the developing infant. We hypothesize that infants with elevated inflammation would also have greater inflammatory immune cell proportions than their formula-fed counterparts.

CONTACTS AND LOCATIONS:
Overall Officials: Bethaney Fehrenkamp, PhD, Principal Investigator — University of Idaho Clinical Assistant Professor
Locations (1):
- University of Idaho, Moscow, Idaho, United States

IPD SHARING:
Plan to Share IPD: No
Only deidentified data or samples will be shared with other researchers. The PI will ensure data confidentiality and deidentification of all data.